CLINICAL TRIAL: NCT02026310
Title: Efficacy/Safety Study of Adding Glimepiride to Type 2 Diabetes Patients With Inadequate Glycemic Control Based on Combination With Metformin And Basal Insulin
Brief Title: Efficacy/Safety Study of Glimepiride to Type 2 Diabetes Patients Based on Metformin And Basal Insulin Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qifu Li (Other)
Responsible Party: Sponsor-Investigator, Qifu Li, Qifu Li, Chongqing Medical University, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: yml2013
Record Dates: First submitted 2013-12-26; First posted 2014-01-01 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: glimepiride; metformin; basal insulin; Hemoglobin A, Glycosylated; glucose fluctuation; hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia | interventions — glimepiride; Insulin Glargine; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- glimepiride (Experimental): on the basis of metformin and glargine, the initial dose of glimepiride is 2 mg,qd (before breakfast), and adjust the dosage for fasting plasma glucose, dosage-adding indicator is the FPG≥7.2, maximum dose of glimepiride is 4 mg/d per day.
  Interventions: Drug: glimepiride; Drug: glargine and metformin
- Metformin and glargine (Active Comparator): on the basis of Metformin and glargine,no glempiride addition. dose of glargine was adjust according to the FPG, with the target less than 7.2mmol/l
  Interventions: Drug: glargine and metformin

INTERVENTIONS:
Drug: glimepiride — on the basis of metformin and glargine, glimepiride is added; with the maximun dose of glimepiride, if the targeted FPG is not reached, glargine dose will be increased.
  Arms: glimepiride
Drug: glargine and metformin
  Other Names: lantus

SUMMARY:
All the guidelines suggest that metformin as the basis of type 2 diabetes medication, and evidence is sufficient.At the same time the basal insulin injection once a day are more and more widely used in diabetes patients in China.

This study aims to evaluate the efficacy and safety of adding glimepiride to type 2 diabetes patients with inadequate glycemic control with combined therapy of metformin and basal insulin.

ELIGIBILITY:
Inclusion Criteria:

* Understand the whole test process, voluntary and signed informed consent form
* Men and women aged 35 to 70 years old
* 20≤BMI<35 Kg/m2
* Diagnosed with type 2 diabetes
* Undergoing metformin(Dose not less than 1000 mg/day)in combination with basal insulin injection once a day
* HbA1c7.0-11%
* Patients should be able to self blood glucose monitoring

Exclusion Criteria:

* sulfonylureas,glinides,TZDs use within 3 months before the study
* Pregnant or lactating women
* A history of ketoacidosis
* Allergy to sulfonylureas or sulfa drug patients
* Apparent dysfunction of liver and kidney patients(ALT>2 times upper normal limit,serum creatinine>1.2 times upper normal limit)
* Poor blood pressure control(systolic pressure>180mmHg or diastolic blood pressure>110mmHg)
* heart disease,cardiac insufficiency,unstable angina pectoris,ECG indicates left ventricle hypertrophy,severe anemia(Hb<9.0g/d1)
* Severe diabetic nerve complications(ulcer of lower limb,neurogenic bladder)
* BMI<20 orBMI≥35kg/m2
* Alcohol or drug abuse ,or can't collaborate due to mental disorder
* Digestion and absorption function obstacle or Other endocrine disorders
* Other chronic diseases required long-term glucocorticoid treatment

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
24 weeks after treatment, HbA1c values' change compared with baseline | 24 weeks after treatment

SECONDARY OUTCOMES:
hypoglycemia events | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Li Qifu, PhD, Study Chair — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Yang W, Lu J, Weng J, Jia W, Ji L, Xiao J, Shan Z, Liu J, Tian H, Ji Q, Zhu D, Ge J, Lin L, Chen L, Guo X, Zhao Z, Li Q, Zhou Z, Shan G, He J; China National Diabetes and Metabolic Disorders Study Group. Prevalence of diabetes among men and women in China. N Engl J Med. 2010 Mar 25;362(12):1090-101. doi: 10.1056/NEJMoa0908292. PMID 20335585
- [Background] Abdul-Ghani MA, DeFronzo RA. Pathogenesis of insulin resistance in skeletal muscle. J Biomed Biotechnol. 2010;2010:476279. doi: 10.1155/2010/476279. Epub 2010 Apr 26. PMID 20445742
- [Background] Holman RR, Paul SK, Bethel MA, Matthews DR, Neil HA. 10-year follow-up of intensive glucose control in type 2 diabetes. N Engl J Med. 2008 Oct 9;359(15):1577-89. doi: 10.1056/NEJMoa0806470. Epub 2008 Sep 10. PMID 18784090
- [Background] Yki-Jarvinen H, Ryysy L, Nikkila K, Tulokas T, Vanamo R, Heikkila M. Comparison of bedtime insulin regimens in patients with type 2 diabetes mellitus. A randomized, controlled trial. Ann Intern Med. 1999 Mar 2;130(5):389-96. doi: 10.7326/0003-4819-130-5-199903020-00002. PMID 10068412
- [Background] Overkamp D, Volk A, Maerker E, Heide PE, Wahl HG, Rett K, Haring HU. Acute effect of glimepiride on insulin-stimulated glucose metabolism in glucose-tolerant insulin-resistant offspring of patients with type 2 diabetes. Diabetes Care. 2002 Nov;25(11):2065-73. doi: 10.2337/diacare.25.11.2065. PMID 12401758